CLINICAL TRIAL: NCT07105982
Title: Clinical Application of a Novel Radiolabeled Translocator Protein (TSPO) Targeted Small Molecular Probe in Inflammation Imaging of Acute Myocardial Infarction
Brief Title: Radiolabeled TSPO Targeted Molecular Probe in AMI
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Feng Wang, Chief physician, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20250624-07-KS-01
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Acute Myocardial Infarction (AMI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the clinical application value of the novel radiolabeled TSPO-targeted molecular probe Gallium [68Ga]-DOTA-HK-011 for inflammation imaging associated with acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers, patients, or their legal representatives must sign the informed consent form and be able to cooperate with the PET-MR examination by lying flat for more than 30 minutes and maintaining a stable position.
* No gender restrictions; age between 18 and 75 years, inclusive.
* Patients must meet the diagnostic criteria for acute myocardial infarction (AMI), such as elevated myocardial enzyme spectrum, dynamic changes in electrocardiogram, or confirmation by coronary angiography.
* Patients who are 7 to 10 days post-onset of acute myocardial infarction.
* Renal GFR > 50 ml/min; ERPF > 280 ml/min; platelet count (PLT) > 75,000/μL; white blood cells (WBC) > 3,000/μL; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels less than three times the upper limit of normal.

Exclusion Criteria:

* Individuals with a history of allergy to similar drugs (drugs with similar chemical or biological components to TSPO), a history of allergies, or currently suffering from allergic diseases.
* Use of anti-inflammatory drugs (such as corticosteroids or immunosuppressants) within the last 14 days, which may affect inflammation imaging.
* Hemodynamically unstable conditions (such as cardiogenic shock or severe arrhythmias); Recent cerebral hemorrhage or severe bleeding tendency within the last 30 days.
* Red blood cell count (RBC) < 4×10^12/L, white blood cell count (WBC) < 3×10^9/L, hemoglobin less than 110 g/L, platelet count (PLT) < 75×10^9/L.
* Significant abnormal liver or kidney function, with glomerular filtration rate (GFR) less than 50 ml/min.
* Presence of ferromagnetic metals implanted in the body (such as cardiac pacemakers, artificial heart valves, metal stents, etc.).
* Claustrophobia or inability to tolerate prolonged examinations.
* Presence of severe acute concomitant diseases or severe refractory mental disorders.
* Pregnant or breastfeeding women (pregnancy defined as a positive urine pregnancy test).
* Patients whose physical condition contraindicates radioactive examinations, such as severe cardiopulmonary insufficiency or other conditions deemed unsuitable by the investigator.
* Other circumstances deemed unsuitable for participation in the trial by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited through hospital electronic records and community health centers
Sampling Method: Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax of lesion uptake value | Time Frame: 60min after administration